CLINICAL TRIAL: NCT07147777
Title: Effect of Physical Activity During Pregnancy on Uterine Artery Blood Flow, Fetal Heart Rate and Fetal Birth Weight
Brief Title: The Effect of Physical Activity During Pregnancy on Uterine and Fetal Parameters
Acronym: TEOPADPUFP
Status: Completed | Type: Observational
Sponsor: Antalya Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: Antalya City/Anatolian Hosp
Record Dates: First submitted 2025-08-22; First posted 2025-08-29 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Pregnancy; Physical Activity
Keywords: pregnancy; physical activity; PPAQ; uterine blood flow; fetal heart rate; birth weight
MeSH Terms: conditions — Motor Activity; Birth Weight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Inactive group: Pregnant women will be divided into three categories based on the distribution of their PPAQ scores: the bottom 33% (inactive group), the middle 33% (moderately active group), and the top 33% (overactive group).
- Moderately active group: Pregnant women will be divided into three categories based on the distribution of their PPAQ scores: the bottom 33% (inactive group), the middle 33% (moderately active group), and the top 33% (overactive group).
- Overactive group: Pregnant women will be divided into three categories based on the distribution of their PPAQ scores: the bottom 33% (inactive group), the middle 33% (moderately active group), and the top 33% (overactive group).

SUMMARY:
This study investigates the relationship between physical activity levels and fetal health in the third trimester of pregnancy. Using the PPAQ and daily step counts, researchers will measure physical activity and examine its effects on uterine blood flow, fetal heart rate, and birth weight. The study hypothesizes that both inactivity and excessive activity may negatively impact fetal health. By focusing on overall activity levels rather than acute effects, this research aims to provide new insights to inform recommendations for a healthy pregnancy.

DETAILED DESCRIPTION:
Urbanization, rising living standards, and the comfort afforded by technological advances, characteristic of our age, are leading to the prevalence of physical inactivity. The potential effects of this on maternal and fetal health, especially during a sensitive period like pregnancy, pose a critical need for scientific research. The third trimester of pregnancy is a critical period during which fetal growth and development occur rapidly, and investigating the effects of physical inactivity on the fetus is of great importance.

In this study, physical activity levels during pregnancy will be determined using the Pregnancy Physical Activity Questionnaire (PPAQ) and daily step count. Fetal health parameters will include uterine blood flow markers (Resistance Index (RI), Systolic/Diastolic (S/D) ratio), fetal heart rate, and fetal birth weight. This study aims to make significant contributions to the literature by revealing the impact of physical activity levels on fetal health parameters in third-trimester pregnancies. Research Hypothesis:

This study will examine the effects of physical activity levels on fetal health parameters within the framework of the following hypotheses:

H1 (Research Hypothesis 1): It is hypothesized that fetal health parameters will be negatively affected in pregnant women who are physically inactive during pregnancy (e.g., impaired values, low birth weight).

H0 (Null Hypothesis 1): There is no statistically significant difference in fetal health parameters between pregnant women who are physically inactive during pregnancy and those who are active.

H2 (Research Hypothesis 2): It is hypothesized that fetal health parameters may also be negatively affected in pregnant women who are excessively physically active during pregnancy (e.g., impaired values, low birth weight), and that there is an optimal physical activity level for pregnancy.

H0 (Null Hypothesis 2): There is no linear relationship between physical activity levels during pregnancy and fetal heart rate and fetal health parameters, and excessive physical activity does not have a negative effect on these parameters. No specific studies have been found examining the relationship between physical activity level measured with the PPAQ and phone step count in the last trimester of pregnancy and uterine artery blood flow, fetal heart rate, and fetal birth weight. However, there are related research themes:

A study by Nguyen et al. found that moderate-intensity recreational physical activity was associated with a higher uterine artery pulsatility index and an increased risk of uterine artery notching. Conversely, moderate-intensity work activity was associated with a lower uterine artery pulsatility index and a reduced risk of uterine artery notching. No association was found with umbilical circulation (1). A study measured uterine artery blood flow in pregnant women and investigated its relationship with the mother's physical fitness level. This study showed that moderate, regular physical activity or inactivity in mothers during pregnancy did not affect resting uterine artery blood flow. In other words, no direct link has been found between the mother's physical fitness level and uterine blood flow. A randomized controlled trial on pregnancy activity examined the longitudinal effects of a supervised, moderate-intensity exercise program on uterine-placental and fetal blood flow parameters. The study observed no deterioration in fetal or maternal Doppler parameters in the exercise group. This suggests that the baby's health is not adversely affected by exercise.

A review on this topic has indicated that exercise during pregnancy can cause a temporary and harmless increase in fetal heart rate, which quickly returns to normal. It has also been revealed that uterine blood flow may decrease partially during exercise, but this is compensated for by physiological adaptations in the mother and quickly returns to normal, with little or no effect on fetal blood flow. The effects on birth weight vary across studies: some studies suggest that exercise may lead to lower birth weight, while others suggest no difference or that moderate-intensity exercise may have positive effects. This review emphasizes that strenuous exercise may increase the risk of low birth weight.

Furthermore, according to this review, if there are no obstetric or medical risks associated with exercise, pregnant women should be encouraged to engage in regular, moderate-intensity exercise programs. Beneficial exercises during pregnancy include walking, running/treadmill exercises, aerobics, swimming, and yoga. Extremely challenging sports and rapid immersion in water are not recommended during pregnancy. Pregnancy is not a prison, and healthy pregnant women should be encouraged to participate in and maintain physical activity.

This study will make a significant and original contribution to the literature because it is one of the first to assess the overall physical activity level of pregnant women, rather than the immediate effects of physical activity, and to measure fetal health parameters such as uterine artery blood flow, fetal heart rate, and fetal birth weight. While most existing research generally focuses on the short-term or acute effects of physical activity, this study aims to provide a more long-term and comprehensive analysis. In this context, physical activity level will be determined by Metabolic Equivalent of Task (MET) obtained through the Pregnancy Physical Activity Questionnaire (PPAQ). MET is a standard unit of measurement that indicates how much energy an activity expends compared to rest. Additionally, average step count data obtained from smartphones and watches will be used to assess overall physical activity levels.

Objective measurements of uterine artery blood flow will be made in the study. These measurements include parameters such as RI, which reflects blood flow resistance in the vessels. RI is the difference between systolic and diastolic velocity divided by systolic velocity. The S/D ratio will also be examined. Combining all these Doppler measurements with objective measurements such as fetal heart rate and birth weight will significantly increase the scientific value of the study.

The primary objective of this study is to determine the potential effects of a sedentary lifestyle on fetal health during the third trimester of pregnancy. This will contribute to the development of more informed recommendations for activity during pregnancy and the protection of maternal and fetal health. The data obtained will provide a scientific basis for healthcare professionals to better guide their clients.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* ≥28 gestational weeks (confirmed by ultrasound)
* Willing and able to participate; provides written informed consent
* Owns a mobile phone capable of step-count data collection

Exclusion Criteria:

* Multiple pregnancy
* History of miscarriage in previous pregnancies
* Chronic systemic disease (e.g., diabetes, hypertension, thyroid disease)
* Detection of fetal anomalies
* Drug or substance abuse
* Current cigarette smoking
* Serious psychiatric illness

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Study participants are limited to pregnant women, which requires female biological sex.
Study Population: Patients were selected by systematic random sampling method among pregnant women who applied to the obstetrics clinic and were in the last trimester of their pregnancy (28th week and following weeks).
Sampling Method: Probability Sample
Enrollment: 159 (Actual)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-12-15 (Actual)

PRIMARY OUTCOMES:
Resistance index measurement | 28-40 weeks of gestation
  Systolic speed minus diastolic speed divided by systolic speed
Systolic-diastolic ratio measurement | 28-40 weeks of gestation
  Systolic value divided by diastolic value on ultrasound
Fetal hearth rate measurement | 28-40 weeks of gestation
  Fetal heart rate measured during sonographic obstetric evaluation of the fetus

SECONDARY OUTCOMES:
Baby's birth weight measurement | Day of delivery
  The baby's first weight measured in the delivery room

CONTACTS AND LOCATIONS:
Overall Officials: Erhan Muluk, MD, Study Chair — Antalya Anatolia Hospital
Locations (1):
- Antalya City Hospital, Antalya Anatolia Hospital, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The de-identified individual participant data (IPD) from this study, along with the study protocol and statistical analysis plan, will be made available to researchers who provide a methodologically sound proposal. The data will be shared after publication of the main results, through a secure platform, for a period of up to 5 years.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 5 years
Access Criteria: De-identified individual participant data will be made available to researchers who provide a methodologically sound and ethically approved research proposal. Data will be shared via a secure, designated platform, and a data use agreement will be required to ensure compliance with privacy and ethical standards.
URL: https://zenodo.org/records/16928837

REFERENCES:
- [Background] Köken G, Yılmazer M. Gebelik ve Egzersiz. Turkiye Klinikleri J Gynecol Obst. 2007;17:385-92.
- [Background] Shanklin DR. Letter to editor revised. N Engl J Med. 1973 Aug 2;289(5):273-4. doi: 10.1056/NEJM197308022890521. No abstract available. PMID 4713775
- [Background] Park S, Marcotte R, Staudenmayer J, Sirard J, VanKim N, Pekow P, Strath S, Freedson P, Chasan-Taber L. Validity of the Pregnancy Physical Activity Questionnaire Short Form (PPAQ-SF). Am J Epidemiol. 2024 Oct 2:kwae382. doi: 10.1093/aje/kwae382. Online ahead of print. PMID 39359005
- [Background] Fernandez-Buhigas I, Martin Arias A, Vargas-Terrones M, Brik M, Rolle V, Barakat R, Munoz-Gonzalez MD, Refoyo I, Gil MM, Santacruz B. Fetal and maternal Doppler adaptation to maternal exercise during pregnancy: a randomized controlled trial. J Matern Fetal Neonatal Med. 2023 Dec;36(1):2183759. doi: 10.1080/14767058.2023.2183759. PMID 36889747
- [Background] Sussman D, Saini BS, Schneiderman JE, Spitzer R, Seed M, Lye SJ, Wells GD. Uterine artery and umbilical vein blood flow are unaffected by moderate habitual physical activity during pregnancy. Prenat Diagn. 2019 Oct;39(11):976-985. doi: 10.1002/pd.5517. Epub 2019 Jul 29. PMID 31254464
- [Background] Nguyen NC, Evenson KR, Savitz DA, Chu H, Thorp JM, Daniels JL. Physical activity and maternal-fetal circulation measured by Doppler ultrasound. J Perinatol. 2013 Feb;33(2):87-93. doi: 10.1038/jp.2012.68. Epub 2012 Jun 7. PMID 22678142